CLINICAL TRIAL: NCT05225090
Title: Trial of a Smartphone Application to Improve Medication Adherence Among Patients with Cancer
Brief Title: Smartphone App for Cancer Medication Adherence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Melissa K Accordino, Assistant Professor of Medicine, Division of Hematology/Oncology, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: AAAS5950
Record Dates: First submitted 2021-03-11; First posted 2022-02-04 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Carcinoma; Cancer
Keywords: any stage
MeSH Terms: conditions — Carcinoma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Smartphone App Intervention (Other): Cancer patients taking at least one oral anti-cancer drug or oral medication to manage a chronic condition in conjunction with any cancer treatment will receive messages through the Medisafe App.
  Interventions: Other: Smartphone App

INTERVENTIONS:
Other: Smartphone App — Medisafe is a Med_App that is free and has been used in several studies evaluating medication adherence. Patients will receive individualized instruction and be followed for 12 weeks. The researcher will show the patients how to input current medication list, set up medication reminders and track if daily doses have been taken using the App (20 minute training session). After the participant has input their medication information into the app, the researcher will assist the participant in adding an optional "Medifriend" who will be alerted if the participant misses a dose as an option. The participant will also be provided with written instructions about the Medisafe app to take home for reference. At each office visit (4, 8, and 12 weeks) participants will complete a medication checklist and reconciliation form with the research staff. Participants will also be asked to send a medication status report through the Medisafe app.
  Other Names: Medisafe App

SUMMARY:
For this current proposal, the investigator will conduct a single-center prospective non-randomized pilot interventional study in patients with any stage and type of cancer who are either taking at least one OACD or are taking at least one oral medication for chronic condition management in conjunction with any cancer treatment.

Primary Objective: To determine the feasibility of using a medication reminder application (Medisafe App) to improve medication adherence in cancer patients either receiving oral anticancer agents (OACDs) or receiving oral medications for chronic disease management (non-OACDs) in conjunction with non-oral cancer treatment.

Secondary Objectives: To compare and characterize medication adherence before and after the 12-week intervention using the Voils Extent of Adherence Scale and the Medisafe App. Also to determine the acceptability, utility and patient engagement with the App, to evaluate changes in healthcare related quality of life before and after the intervention, and to explore behaviors, knowledge, attitudes and beliefs related to medication adherence using a semi-structured interview delivered over the telephone.

DETAILED DESCRIPTION:
Many patients with cancer experience frustration with the large number and complex scheduling of their medications. This study will help find out how much "pill burden" exists in patients with cancer, and how a smartphone app can help patients take medications as providers prescribe. Results of this study may help figure out the best way to help patients manage medications in the future.

ELIGIBILITY:
Inclusion Criteria:

* Any type/stage cancer
* Patients must be taking either:

  * at least one oral anti-cancer drug (OACD) or
  * at least one oral medication (non-OACD) for management of a chronic condition in addition to receiving non-oral cancer treatment
* Patients must have access to a mobile phone or tablet that can download the Medisafe App. (ie apple/android)
* Subjects must be able to complete self-administered questionnaires in English or Spanish.
* Co-enrollment in trials involving pharmacologic therapy is allowed.

Exclusion Criteria:

* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects enrolled that complete the 12-week intervention and assessments | 12 weeks
  To determine the feasibility of using a medication reminder application (Medisafe App) to improve medication adherence in cancer patients. Feasibility defined as completing the 12-week intervention and the endpoint assessments. Patients will be tallied.

SECONDARY OUTCOMES:
Change in mean score on the Voils Extent of Adherence Scale for oral caner therapy use between baseline and 12 weeks | Baseline and 12 weeks
  To compare medical adherence to OACDs before and after the 12-week intervention using the Voils Extent of Adherence Scale for OACD use. The Extent of Adherence subscale of the Voils Self-Reported Medication Nonadherence Measurement (Voils Measure) will be used for self-assessment of drug adherence. The Extent of Adherence subscale of the Voils Measure consists of three questions with responses ranging from 1 (perfect adherence) to 5 (highest degree of nonadherence). The Extent score can be calculated in two different ways: the three items in the Extent scale can be averaged, with higher scores representing greater nonadherence, or the scale can be dichotomized, such that perfect adherence is considered "adherent", and any degree of nonadherence is considered "nonadherent."
Change in mean score on the Voils Extent of Adherence Scale for global medication use between baseline and 12 weeks | Baseline and 12 weeks
  To compare medical adherence to OACDs before and after the 12-week intervention using the Voils Extent of Adherence Scale for OACD use. The Extent of Adherence subscale of the Voils Self-Reported Medication Nonadherence Measurement (Voils Measure) will be used for self-assessment of drug adherence. The Extent of Adherence subscale of the Voils Measure consists of three questions with responses ranging from 1 (perfect adherence) to 5 (highest degree of nonadherence). The Extent score can be calculated in two different ways: the three items in the Extent scale can be averaged, with higher scores representing greater nonadherence, or the scale can be dichotomized, such that perfect adherence is considered "adherent", and any degree of nonadherence is considered "nonadherent." For this study, global adherence will be defined as a perfect score (1) for each medication.
Mean Score to Medication Self-Efficacy Scale (MASES) to assess a patient's confidence in their ability to take their medications in a variety of situations | 12 weeks
  The Medication Self-Efficacy Scale (MASES) is a tool used to assess a patient's confidence in their ability to take their medications in a variety of situations. This is a 25-item scale and items are scored 1= not sure at all, to 4= very sure, and the total scores of the measure is the mean response to all the items (range 1-4).
Mean Score on the User Version of the Mobile Application Rating Scale | 12 weeks
  The User Version of the Mobile Application Rating Scale (uMARS) is a 20-item tool used for classifying and assessing the quality of mobile health apps. It contains four objective quality subscales including engagement, functionality, aesthetics, and information quality. Each of the 20-items have an outcome of 1-5; the overall outcome scale ranges from 20-100. It has been developed and validated specifically for end user administration.
Change in Patient-Reported Outcomes Measurement Information System (PROMIS) 29 Score before and after the intervention | Baseline and 12 weeks
  The Patient-Reported Outcomes Measurement Information System (PROMIS) 29 is a well- validated assessment tool that offers both qualitative and quantitative measures of health-related quality of life. The PROMIS-29 includes 29 questions evaluating areas of physical function, anxiety, depression, fatigue, sleep, social functioning, and pain interference. The PROMIS-29 assesses severity levels of symptoms and their effect on the patient's functioning.
Change in Treatment Satisfaction Questionnaire for Medication (TSQM) Domain Score before and after the intervention | Baseline and 12 weeks
  The 14-item TSQM Version 1.4 is a reliable and valid instrument to assess patients' satisfaction with medication, providing scores on four scales - side effects, effectiveness, convenience and global satisfaction. We will use the validated abbreviated TSQM-9.24 This questionnaire includes 9-items that address six different domains which include domains of TS-M included; (1) side effects, (2) symptom relief, (3) convenience, (4) effectiveness, (5) impact on daily life, and (6) tolerability/acceptability. Scoring of the TSQM-9 provides a domain score that ranges from 0- 100 with higher scores representing higher satisfaction on each domain.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Accordino, MD, Principal Investigator — Assistant Professor of Medicine
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No